CLINICAL TRIAL: NCT03727984
Title: Demographic, Clinical Characteristics and Medications of Re-hospitalized Patients for Acute Coronary Syndrome
Brief Title: Re-hospitalized Patients With Acute Coronary Syndrome
Acronym: BoomerangACS
Status: Completed | Type: Observational
Sponsor: Cardiovascular Academy Society, Turkey (Other)
Responsible Party: Principal Investigator, Mehdi Zoghi, Prof. Dr., Cardiovascular Academy Society, Turkey
Other Study IDs: 2018-2
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Myocardial infarction; Hospitalization; Coronary artery disease; Retrospective; Cohort study
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The predictors of re-hospitalization of patients with history of acute coronary syndrome

DETAILED DESCRIPTION:
The aim of this retrospective multicenter study is to evaluate the demographic, clinical characteristics and medications of re-hospitalized for new cardiac event in patients with history of acute coronary syndrome within in 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patients age >18 years who had hospitalized for acute coronary syndrome within 12 months

Exclusion Criteria:

Patients whose previous hospitalizations data are not available Myocardial Infarction, type 2 patients

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The aim of this retrospective multicenter study is to evaluate the demographic, clinical characteristics and medications of re-hospitalized for new cardiac event in patients with history of acute coronary syndrome within in 12 months. To the best of our knowledge, this is the first study to evaluate the characteristics of re-hospitalized patients for ACS. The case report forms which attached in excel must be filled by investigators case by case based on recorded data.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Clinical and demographics characteristics of patients re-admitted with acute coronary syndrome | Up to 1 year
  The demographics and clinical characteristics of study population Admissions with an 'I'-group ICD-10 code
Cardiovascular Hospitalization | Up to 1 year
  Predictive factors for patients re-admitted with acute coronary

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Academy Society, Izmir, Turkey (Türkiye)